CLINICAL TRIAL: NCT06535880
Title: Brainstem Mapping of Nociceptive and Non-nociceptive Trigeminal Input and Its Functional Connectivty
Brief Title: Trigeminal Brainstem Mapping 2: Higher Cortical Strucureas As Well As Subnuclei of the Spinal Trigeminal Nucleus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TrigeminalBrainstemMapping2
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electric Stimulation (Experimental): Electric stimulation with a Digitimer DS7AH HV Current Stimulator delivered with 4 shielded electrodes mounted on the participants head and arm.
  Interventions: Device: Electric Current Stimulation

INTERVENTIONS:
Device: Electric Current Stimulation — Electric stimulation with a Digitimer DS7AH HV Current Stimulator delivered with 4 shielded electrodes mounted on the participants head and arm

SUMMARY:
In previous studies clustering of the three branches of the trigeminal nerve in brainstem were shown, cerebellum and periaqueductal gray. To further evaluate higher cortical structures, which were not covered by our previous field of view (FOV) and to further investigate the identified 'subnuclei' of the spinal trigeminal nucleus, here the aim is to scan the whole brain as well as the brainstem and the upper spinal cord during trigeminal nociceptive as well as non-nociceptive electrical stimulation of all three branches of the trigeminal nerve (and the arm as a somatic control site) during acquisition of BOLD-fMRI in humans.

DETAILED DESCRIPTION:
Preprocessing and processing of the MR data will follow our previous publications (Mehnert et al 2023, Mehnert et al 2024)

ELIGIBILITY:
Inclusion Criteria:

* healthy
* suitable fo MRI

Exclusion Criteria:

* headache disease
* psychological disorder
* pregnancy
* all exclusion criteria necessary for imaging in a 3 T MRI scanner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Statistical Parametric Maps calculated from the fMRI data on brainstem level | only 1 visit
  At an small volume corrected threshold of p<0.05 will be reproduce activation of all previously shown subnuclei of the spinal trigeminal nucleus for all three trigeminal branches using a sphere of 10 mm around previously published (Mehnert et al, 2023) MNI coordinates.
Statistical Parametric Maps calculated from the fMRI data of higher cortical brain structures | only 1 visit
  Anterior and posterior insula, the cingulate cortex and S1/S2 will show significant activation at an small-volume corrected threshold of p<0.05

SECONDARY OUTCOMES:
Functional connectivty between insula and spinal trigeminal cortex | only 1 visit
  For each of the trigeminal subnuclei we will calculate the functional connectivity to higher cortical areas, such as the anterior and posterior insula, the cingulate cortex and S1/S2 with a psycho-physiological interaction analysis (PPI) for painful as well as non-painful stimulation to characterize the function of each subnucleus.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehnert J, Basedau H, Sturm LM, Nielsen T, Jensen RH, May A. Functional brainstem representations of the human trigeminal cervical complex. Cephalalgia. 2023 May;43(5):3331024231174862. doi: 10.1177/03331024231174862. PMID 37203351
- [Background] Basedau H, May A, Mehnert J. Cerebellar somatotopy of the trigemino-cervical complex during nociception. Eur J Pain. 2024 May;28(5):719-728. doi: 10.1002/ejp.2212. Epub 2023 Nov 28. PMID 38013614
- [Background] Mehnert J, Tinnermann A, Basedau H, May A. Functional representation of trigeminal nociceptive input in the human periaqueductal gray. Sci Adv. 2024 Mar 22;10(12):eadj8213. doi: 10.1126/sciadv.adj8213. Epub 2024 Mar 20. PMID 38507498